CLINICAL TRIAL: NCT03655730
Title: Efficacity of a Sustained Weekly Psychological Intervention for Adolescents and Young Adults Attending to Local Missions for Reinsertion, on Reducing the Suicidal Ideations, Depression Level and Improving Reinsertion Compared to Usual Care
Brief Title: Efficacity of Psychological Intervention on Reducing the Suicidal Ideations, Depression Level and Improving Reinsertion
Acronym: MLADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K170104-J; 2018-A01255-50 (Other: IDRCB)
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Depressive Symptoms
Keywords: Depression; suicidal risk; self-harm behavior; young people
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This study is a comparative, randomised controlled trial that aims at demonstrating the superiority of weekly psychotherapeutic intervention during one year in lowering depression symptoms compared to usual care.
  The ratio between intervention and usual care arms will be 1:1.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): follow weekly psychotherapeutic individual sessions following the IPT method during one year.
  Interventions: Other: weekly psychotherapeutic individual sessions; Other: Usual care
- usual care arm (Experimental): continue with the standard follow-up provided by the Mission Locale, including periodic meetings with a referee
  Interventions: Other: Usual care

INTERVENTIONS:
Other: weekly psychotherapeutic individual sessions — weekly psychotherapeutic individual sessions following the IPT method during one year
  Arms: intervention arm
Other: Usual care — the standard follow-up provided by the Mission Locale, including periodic meetings with a referee

SUMMARY:
Suicide is the third leading cause of death in adolescents and young adults in the United States and the second leading cause in European countries.

Depressive disorders are consistently the most prevalent psychiatric disorder among adolescents who attempt suicide with a prevalence ranging from 49% to 64%. Depression in adolescent and young adults is a multifactorial phenomenon, as is the risk of suicidal attempt. To address such problems, effective and accessible treatment is needed, as recommended by the French Health Authority (HAS).

Our primary objective is to demonstrate that a weekly psychotherapeutic intervention reduces the depression level.

The primary assessment criterion is the variation of the clinician Adolescent Depression Rating Scale (ADRSc) from randomisation to month 6.

The study also aims comparing in the 2 randomised groups

* ADRS depression global score (clinician and subject) at 0, 3, 9 and 12 months
* Number of suicidal attempts and self-harm attempts at 6 and 12 months
* Number of drop-out at 6 and 12 months
* Beck's Hopelessness Scale at 0, 3, 6, 9 and 12 months
* Global score on the GHQ-28 and scores on the 4 subscales (Somatization, Anxiety and Insomnia, Social dysfunction, Depressive mood) at 0, 3, 6, 9 and 12 months.
* Working AIliance Inventory (WAI) score at 0, 3, 6, 9 and 12 months

DETAILED DESCRIPTION:
Suicide is the third leading cause of death in adolescents and young adults in the United States and the second leading cause in European countries. In France, recent epidemiological data showed that the suicide rate in adolescents aged 15 to 19 is 4.1/100 000 inhabitants. Prevalence of suicidal ideations ranges from 15 to 25% in the general population and lifetime estimates of suicide attempts among adolescents range from 1.3 to 3.8% in males and from 1.5 to 10.1% in females. Reducing suicide and suicide attempts is therefore a key public health target.

Depressive disorders are consistently the most prevalent psychiatric disorder among adolescents who attempt suicide with a prevalence ranging from 49% to 64%. Depression in adolescent and young adults is a multifactorial phenomenon, as is the risk of suicidal attempt.

Being in a situation of failure at school or not having a clear training or work project clearly increases the risk for depression. Some studies have targeted potential high school drop outs as a target for prevention of suicidality.

To address such problems, effective and accessible treatment is needed, as recommended by the French Health Authority (HAS). However, only few studies assess, through a randomized protocol, efficacity and feasibility of psychotherapeutic treatment in psychiatry in general and particularly in this population, although individual psychotherapy is highly recommended in clinical practice for depressed adolescents and young adults.

Our primary objective is to demonstrate that a weekly psychotherapeutic intervention reduces the depression level.

The primary assessment criterion is the variation of the clinician Adolescent Depression Rating Scale (ADRSc) from randomisation to month 6.

Others objectives are the following :

To compare in the 2 randomised groups

* ADRS depression global score (clinician and subject) at 0, 3, 9 and 12 months
* Number of suicidal attempts and self-harm attempts at 6 and 12 months
* Number of drop-out at 6 and 12 months
* Beck's Hopelessness Scale at 0, 3, 6, 9 and 12 months
* Global score on the GHQ-28 and scores on the 4 subscales (Somatization, Anxiety and Insomnia, Social dysfunction, Depressive mood) at 0, 3, 6, 9 and 12 months.
* Working AIliance Inventory (WAI) score at 0, 3, 6, 9 and 12 months

To describe, in the whole sample (randomised and not randomised),

- the baseline level of abuse during childhood with the CTQ. The effectiveness of reinsertion activities (jobs, diploma, attendance to the Mission Locale) at 0, 3, 6, 9 and 12 months

To evaluate the sensitivity to change of the French version of the ADRSc.

330 subjects wil be included to have 132 randomized subjects into two arms: sustained psychotherapeutic intervention or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Be followed in one of the five participating centres of Mission Locale in Paris,
* Be between 16 (inclusive) and 25 (inclusive) years old at the date of inclusion,
* Agrees to participate in the research and, in the case of a minor, the legal representant agrees with the subject's participation in research.
* Have a Social Security number
* Be fluent in French
* With signed informed consent

Exclusion Criteria:

* Be already followed in a mental health/addiction service, attending to a private or public psychiatric service, or abusing drugs.

Randomisation criteria :

Included subjects will be randomised if at least one of the following conditions is met: baseline ADRSc score greater or equal than 8 or abuse and/or deprivation according to the Childhood Trauma Questionnaire (CTQ, short version):

* score greater or equal than 11 relative to physical abuse
* score greater or equal than 16 relative to emotional abuse
* score greater or equal than 14 relative to physical deprivation
* score greater or equal than 11 relative to sexual abuse).

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Depression level | 6 months
  Defined as the difference of ADRS clinician score (cf. Appendix 18.2.1) between inclusion and 6 month.

SECONDARY OUTCOMES:
depression assessed at 0, 3, 9 and 12 months | at 0, 3, 9 and 12 months
  The ADRSc (clinician) questionnaire will be filled out by the assessor at 0, 3 and 9 and 12 months during follow-up visits
suicidal attempts and self-harm attempts | at 6 and 12 months
  The number of suicidal attempts and self-harm attempts, at 6 and 12 months
drop out | at baseline, 6 and 12 months
  The number of drop outs at baseline, 6 and 12 months
time of the hopelessness | t 0, 3, 6, 9 and 12 months
  The evolution on time of the hopelessness, assessed at 0, 3, 6, 9 and 12 months
global score on the GHQ28 | at 0, 3, 6, 9 and 12 months
  5. The evolution on time of the global score on the GHQ28 and on its 4 subscales (Somatization, Anxiety and Insomnia, Social dysfunction, Depressive mood), assessed at 0, 3, 6, 9 and 12 months
working aIliance | at 0, 3, 6, 9 and 12 months
  The evolution on time of the working aIliance at 0, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Guedeney, PhD, Principal Investigator — APHP
Locations (1):
- Bichat hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided